CLINICAL TRIAL: NCT04949347
Title: Glycerin-Preserved, Human-Donor, Corneoscleral Patch Grafts for Glaucoma Drainage Devices
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naris Kitnarong, Associate professor, Siriraj Hospital
Other Study IDs: NK003
Record Dates: First submitted 2019-09-30; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Glaucoma; Graft Failure; Intraocular Pressure
Keywords: glaucoma; glaucoma surgery; patch graft; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glycerin-preserved, human-donor, cornescleral patch grafts: Consecutive glaucoma patients who had undergone glaucoma drainage device implantation using glycerin-preserved, human-donor, cornescleral patch grafts
  Interventions: Biological: glaucoma drainage device implantation

INTERVENTIONS:
Biological: glaucoma drainage device implantation — Glaucoma drainage device implantation, a 350 mm2 Baerveldt (BG 101-350) GDD (Johnson and Johnson, Santa Ana, CA, USA) was performed using glycerin-preserved, human-donor, corneoscleral tissue ( the remaining from a heterologous, human-donor corneal button, obtained from the International Eye Bank of Thailand, after a clear corneal graft had been used for penetrating keratoplasty.) The tissue had been preserved in glycerin using the sterile technique and kept in a medical refrigerator for no longer than 6 months.
  Other Names: glycerine-preserved corneoscleral patch graft

SUMMARY:
This was a retrospective, non-comparative study of 100 eyes of 100 consecutive glaucoma patients who had undergone glaucoma drainage device implantation (Baerveldt shunt) during January 2006 to December 2016. Glycerin-preserved, human-donor, corneoscleral tissue was used as a patch graft to cover the tube portion of the GDD over the sclera. The patch graft related complication was comparable to the previous reports using conventional sclera or pericardium.

DETAILED DESCRIPTION:
This retrospective, non-comparative study was conducted at the Department of Ophthalmology, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand. The medical records of consecutive patients who had undergone glaucoma drainage device implantation employing the fornix-based conjunctival flap technique and using a glycerin-preserved, human-donor, corneoscleral graft. The procedures were carried out by, or under the supervision of, one surgeon (NK) between January 2006 and December 2016 were reviewed. The study protocol was approved by the Siriraj Institutional Review Board, Faculty of Medicine, Siriraj Hospital, Mahidol University.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients who had undergone glaucoma drainage device implantations between January 2006 and December 2016 at Siriraj hospital by or under supervision of one surgeon (NK).
2. The GDD implantation using glycerin-preserved, human-donor, corneoscleral tissue as a patch graft

Exclusion Criteria:

1.Patients who had follow-up period less than 12 months after operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive glaucoma patients who had undergone glaucoma drainage device implantations using glycerin-preserved, human-donor, corneoscleral tissue as a patch graft to cover the tube between January 2006 and December 2016 at Siriraj hospital by or under supervision of one surgeon (NK).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Numbers of eyes with graft related complication | Postoperative period from January 3, 2006 to August 31, 2019
  Numbers of eyes with the patch-graft related complications included tube exposure, infection, leaking, etc

SECONDARY OUTCOMES:
Intraocular pressure | preoperative and postoperative period from January 3, 2006 to August 31, 2019
  The intraocular pressure level (must be less than 21 mmHg.)
numbers of medication | Postoperative period from January 3, 2006 to August 31, 2019
  Numbers of post-operative anti-glaucoma medication comparing to pre-operative medications
Visual acuity | Postoperative period from January 3, 2006 to August 31, 2019
  The level of post-operative visual acuity compared to pre-operative visual acuity
Numbers and types of post-operative intervention | Postoperative period from January 3, 2006 to August 31, 2019
  Numbers and types of post-operative intervention to correct the complication

CONTACTS AND LOCATIONS:
Overall Officials: Naris Kitnarong, M.D., M.B.A., Principal Investigator — Mahidol University
Locations (1):
- Naris Kitnarong, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsoukanas D, Xanthopoulou P, Charonis AC, Theodossiadis P, Kopsinis G, Filippopoulos T. Heterologous, Fresh, Human Donor Sclera as Patch Graft Material in Glaucoma Drainage Device Surgery. J Glaucoma. 2016 Jul;25(7):558-64. doi: 10.1097/IJG.0000000000000294. PMID 26091179
- [Result] Gedde SJ, Feuer WJ, Shi W, Lim KS, Barton K, Goyal S, Ahmed IIK, Brandt J; Primary Tube Versus Trabeculectomy Study Group. Treatment Outcomes in the Primary Tube Versus Trabeculectomy Study after 1 Year of Follow-up. Ophthalmology. 2018 May;125(5):650-663. doi: 10.1016/j.ophtha.2018.02.003. Epub 2018 Feb 21. PMID 29477688